CLINICAL TRIAL: NCT04255004
Title: Autologous Peripheral Blood Mononuclear Cells for Limb Salvage in Diabetic Foot Patients With No-option Critical Limb Ischemia
Brief Title: Autologous Peripheral Blood Mononuclear Cells in Diabetic Foot Patients With No-option Critical Limb Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Alessia Scatena, Principal Investigator, Ospedale San Donato
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MONODIAB-19-01
Record Dates: First submitted 2020-01-25; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Critical Limb Ischemia; Diabetic Foot
Keywords: autologous peripheral blood mononuclear cell, diabetic foot
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: We would enroll a cohort of 38 consecutive diabetic patients with CLI in charge at the Diabetic Foot Unit of the San Donato Hospital in Arezzo or referred from other Italian hospitals, who have no option for revascularization or are not further eligible for revascularization according to ESVS ESC 2017 criteria to undergo PB-MNC implantation. Furthermore, an historical control group, with a 1:1 case-control ratio, will be collected backwards from our records, when PBMNCs cellular therapy was not available in our center, with same no-option CLI diagnosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-PBMNC therapy (Active Comparator): Patients in A-PBMNC therapy are treated with wound bed multiple perilesional and intramuscular injections of PBMNC cells suspension (0.2-0.3cc in boluses). This procedure is repeated on each patient for three times, at intervals of 30-45 days from each other.
  Interventions: Device: Pall Celeris System, point of care device for human cell therapy
- No A-PBMNC therapy (No Intervention): Patients in No A-PBMNC therapy receive only supportive treatment including wound care and pain killer drug.

INTERVENTIONS:
Device: Pall Celeris System, point of care device for human cell therapy — Concentration of PB-MNCs autologous cell therapy was produced by a filtration-based point-of-care device. All the procedures were performed in operatory room with anaesthesiologic support (propofol and/or peripheral block). Blood withdrawal (120 ml) was collected through a peripheral venous access. Blood was loaded, and gravity filtration was allowed to proceed until the upstream side of the filter had no remaining blood; filtration last about 10 minutes. During filtration, MNCs were captured in the filter while plasma, platelets (PLTs) and red blood cells (RBCs) were not retained. Immediately concentrate solution is injected in the perilesional area and intramuscular in the foot and the leg (0.2-0.3cc in boluses) below the knee, at intervals of 1-2 cm and to a mean depth of 1.5-2 cm, using a 21G needle. This procedure is repeated on each patient for three times, at intervals of 30-45 days from each other.
  Arms: A-PBMNC therapy

SUMMARY:
The objective of this trial is to determine whether PBMNCs in diabetic patients with critical, non revascularizable limb ischemia can prevent major amputation and affect mortality and healing.

DETAILED DESCRIPTION:
This is an interventional study with historical control group carried out to assess as primary outcome major amputations, overall mortality, number of healed patients in group of patients who received repetitive intra-muscular implant of PBMNCs (3 times; 4-week interval) in comparison to a historical internal control group with a 1:1 case-control ratio. Secondary outcomes are TCPO2, healing time and rest pain.

No-option critical limb ischaemia is defined by evidence of no run-off pedal vessels, failure after several percutaneous intervention and no longer possible re-intervention, failure after infra-genicular bypass grafting, no-walking capacity with severe comorbidities unfit for surgical or endovascular procedures.

Inclusion criteria are: a) ulcers with inadequate perfusion, as indicated by a transcutaneous oxygen pressure value (TcpO2) <30 mmHg; b) ulcers with grade I or II or III and stage C as defined by the Texas University Classification System or W1,2,3 - I 3 - FI 0,1 as defined by the WiFI Classification System c) not eligible for angioplasty or vascular surgery or following failed revascularization; d) possibility to save foot support.

Exclusion criteria are: a) lesion site above the tibial-tarsal joint; b) moderate or severe infection according by the WiFI classification system; c) NYHA class IV; d) Anemia (Hb<8g/dl); e) coagulation disorder/thrombocytopenia (PLT< 50,000 per microliter); f) active cancer/leukemia or lymphoma hematological disease.

Standard of care in both groups includes: diabetes control maximization by the diabetologist, comprehensive foot assessment by the nurse together with the diabetologist, including determination of vibration perception threshold, 10-g monofilament test and TcpO2 measurement, dressings, off-loading and systemic therapy according to the IWGDF guidelines .

Informed consent for participation in the study during the progress of the clinical trial is obtained from all subjects.

Concentration of PB-MNCs autologous cell therapy is produced by a filtration-based point-of-care device with the intended for use intra-operatively, from 120 mL of anticoagulated blood. All the procedures are performed in operatory room with anaesthesiologic support (propofol and/or peripheral block). Blood withdrawal (120 ml) is collected through a peripheral venous access, than loaded and gravity filtration is allowed in about 10 minutes. During filtration, MNCs are captured in the filter while plasma, platelets (PLTs) and red blood cells (RBCs) are not retained. After appropriate surgical debridement of the wound bed multiple perilesional and intramuscular injections of PBMNC cells suspension (0.2-0.3cc in boluses) are injected along the relevant axis below the knee, at intervals of 1-2 cm and to a mean depth of 1.5-2 cm, using a 21G needle. This procedure is repeated on each patient for three times, at intervals of 30-45 days from each other.

Foot-sparing surgery, the removal of all the unviable tissue and the reconstruction of the foot to allow a functional deambulation,is performed at the same time of the last implant in the patients with increased TcpO2 value above 30 mmHg. Between the implants, diabetologists together with nurses evaluated changing in pain, infection signs, wound size, demarcation of the necrosis, granulation tissue formation, perilesional tissue trophism and TcpO2 value to optimize standard of care. After the first treatment, a two years follow-up is registered, with evaluation at 1-3-6-12-18-24 months.

A baseline assessment is carried out, in order to estimate any differences among cases and controls before the treatment. Statistical evaluation includes non-parametric tests (Mann-Whitney U test for independent samples for continuous variables and Cochrane chi-square test for discrete variables), evaluation of Relative Risk (RR), Absolute Risk Reduction (ARR), Relative Risk Reduction (RRR) and Number Needed to Treat (NNT), multivariate survival analysis (Kaplan-Meier's survival analysis model).

ELIGIBILITY:
Inclusion Criteria:

* ulcers with inadequate perfusion, as indicated by a transcutaneous oxygen pressure value (TcpO2) <30 mmHg;
* ulcers with grade I or II or III and stage C as defined by the Texas University Classification System or W1,2,3 - I 3 - FI 0,1 as defined by the WiFI Classification System
* not eligible for angioplasty or vascular surgery or following failed revascularization;
* possibility to save foot support.

Exclusion Criteria:

* lesion site above the tibial-tarsal joint;
* moderate or severe infection according by the WiFI classification system;
* NYHA class IV; d) Anemia (Hb<8g/dl);
* coagulation disorder/thrombocytopenia (PLT< 50,000 per microliter);
* active cancer/leukemia or lymphoma hematological disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Amputation-free survival at 1 month | 1 month
  rate of non amputated limb 1 month after the intervention
Amputation-free survival at 3 months | 3 months
  rate of non amputated limb 3 months after the intervention
Amputation-free survival at 6 months | 6 months
  rate of non amputated limb 6 months after the intervention
Amputation-free survival at 12 months | 12 months
  rate of non amputated limb 12 months after the intervention
Amputation-free survival at 18 months | 18 months
  rate of non amputated limb 18 months after the intervention
Amputation-free survival at 24 months | 24 months
  rate of non amputated limb 24 months after the intervention
risk of death at 1 month | 1 month
  rate of dead subjects 1 month after the intervention
risk of death at 3 months | 3 months
  rate of dead subjects 3 months after the intervention
risk of death at 6 months | 6 months
  rate of dead subjects 6 months after the intervention
risk of death at 12 months | 12 months
  rate of dead subjects 12 months after the intervention
risk of death at 18 months | 18 months
  rate of dead subjects 18 months after the intervention
risk of death at 24 months | 24 months
  rate of dead subjects 24 months after the intervention
probability of healing at 1 month | 1 month
  rate of healed subjects 1 month after the intervention
probability of healing at 3 months | 3 months
  rate of healed subjects 3 months after the intervention
probability of healing at 6 months | 6 months
  rate of healed subjects 6 months after the intervention
probability of healing at 12 months | 12 months
  rate of healed subjects 12 months after the intervention
probability of healing at 18 months | 18 months
  rate of healed subjects 18 months after the intervention
probability of healing at 24 months | 24 months
  rate of healed subjects 24 months after the intervention

SECONDARY OUTCOMES:
transcutaneous oxygen measurement (TcPO2) variation | 0-3 months
  comparison of TcPO2 at the second follow up (3 months after intervention) with the baseline measure
Healing time | within 24 months
  time to reach complete epithelialization
rest pain | 0-1-3 months
  comparison of rest pain measured by a numeric rating scale (NRS) min 0 - max 10, where 10 is the worst pain the patient has felt

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Ercolini, MD, Study Chair — Vascular Surgery Unit San Donato Hospital Arezzo

IPD SHARING:
Plan to Share IPD: No
data should not be shared before study completion and approvation by all the collaborators. Sharing data before this time would jeopardize the integrity of the clinical trial process and risk the scientific validity of the results.

REFERENCES:
- [Background] Abu Dabrh AM, Steffen MW, Undavalli C, Asi N, Wang Z, Elamin MB, Conte MS, Murad MH. The natural history of untreated severe or critical limb ischemia. J Vasc Surg. 2015 Dec;62(6):1642-51.e3. doi: 10.1016/j.jvs.2015.07.065. Epub 2015 Sep 26. PMID 26391460
- [Background] Golomb BA, Dang TT, Criqui MH. Peripheral arterial disease: morbidity and mortality implications. Circulation. 2006 Aug 15;114(7):688-99. doi: 10.1161/CIRCULATIONAHA.105.593442. No abstract available. PMID 16908785
- [Background] Rigato M, Monami M, Fadini GP. Autologous Cell Therapy for Peripheral Arterial Disease: Systematic Review and Meta-Analysis of Randomized, Nonrandomized, and Noncontrolled Studies. Circ Res. 2017 Apr 14;120(8):1326-1340. doi: 10.1161/CIRCRESAHA.116.309045. Epub 2017 Jan 17. PMID 28096194
- [Background] Fantin A, Vieira JM, Gestri G, Denti L, Schwarz Q, Prykhozhij S, Peri F, Wilson SW, Ruhrberg C. Tissue macrophages act as cellular chaperones for vascular anastomosis downstream of VEGF-mediated endothelial tip cell induction. Blood. 2010 Aug 5;116(5):829-40. doi: 10.1182/blood-2009-12-257832. Epub 2010 Apr 19. PMID 20404134
- [Background] Baer C, Squadrito ML, Iruela-Arispe ML, De Palma M. Reciprocal interactions between endothelial cells and macrophages in angiogenic vascular niches. Exp Cell Res. 2013 Jul 1;319(11):1626-34. doi: 10.1016/j.yexcr.2013.03.026. Epub 2013 Mar 28. PMID 23542777
- [Background] Wynn TA, Vannella KM. Macrophages in Tissue Repair, Regeneration, and Fibrosis. Immunity. 2016 Mar 15;44(3):450-462. doi: 10.1016/j.immuni.2016.02.015. PMID 26982353
- [Background] Krzyszczyk P, Schloss R, Palmer A, Berthiaume F. The Role of Macrophages in Acute and Chronic Wound Healing and Interventions to Promote Pro-wound Healing Phenotypes. Front Physiol. 2018 May 1;9:419. doi: 10.3389/fphys.2018.00419. eCollection 2018. PMID 29765329
- [Background] Awad O, Dedkov EI, Jiao C, Bloomer S, Tomanek RJ, Schatteman GC. Differential healing activities of CD34+ and CD14+ endothelial cell progenitors. Arterioscler Thromb Vasc Biol. 2006 Apr;26(4):758-64. doi: 10.1161/01.ATV.0000203513.29227.6f. Epub 2006 Jan 12. PMID 16410458
- [Background] Jarajapu YP, Hazra S, Segal M, Li Calzi S, Jadhao C, Qian K, Mitter SK, Raizada MK, Boulton ME, Grant MB. Vasoreparative dysfunction of CD34+ cells in diabetic individuals involves hypoxic desensitization and impaired autocrine/paracrine mechanisms. PLoS One. 2014 Apr 8;9(4):e93965. doi: 10.1371/journal.pone.0093965. eCollection 2014. PMID 24713821
- [Background] Spaltro G, Straino S, Gambini E, Bassetti B, Persico L, Zoli S, Zanobini M, Capogrossi MC, Spirito R, Quarti C, Pompilio G. Characterization of the Pall Celeris system as a point-of-care device for therapeutic angiogenesis. Cytotherapy. 2015 Sep;17(9):1302-13. doi: 10.1016/j.jcyt.2015.04.006. Epub 2015 May 30. PMID 26038175
- [Background] Moriya J, Minamino T, Tateno K, Shimizu N, Kuwabara Y, Sato Y, Saito Y, Komuro I. Long-term outcome of therapeutic neovascularization using peripheral blood mononuclear cells for limb ischemia. Circ Cardiovasc Interv. 2009 Jun;2(3):245-54. doi: 10.1161/CIRCINTERVENTIONS.108.799361. Epub 2009 Mar 30. PMID 20031722
- [Background] Persiani F, Paolini A, Camilli D, Mascellari L, Platone A, Magenta A, Furgiuele S. Peripheral Blood Mononuclear Cells Therapy for Treatment of Lower Limb Ischemia in Diabetic Patients: A Single-Center Experience. Ann Vasc Surg. 2018 Nov;53:190-196. doi: 10.1016/j.avsg.2018.05.036. Epub 2018 Jul 25. PMID 30053546
- [Background] Armstrong DG, Lavery LA, Harkless LB. Validation of a diabetic wound classification system. The contribution of depth, infection, and ischemia to risk of amputation. Diabetes Care. 1998 May;21(5):855-9. doi: 10.2337/diacare.21.5.855. PMID 9589255
- [Background] Wagner FW Jr. The dysvascular foot: a system for diagnosis and treatment. Foot Ankle. 1981 Sep;2(2):64-122. doi: 10.1177/107110078100200202. No abstract available. PMID 7319435
- [Background] Lipsky BA, Aragon-Sanchez J, Diggle M, Embil J, Kono S, Lavery L, Senneville E, Urbancic-Rovan V, Van Asten S; International Working Group on the Diabetic Foot; Peters EJ. IWGDF guidance on the diagnosis and management of foot infections in persons with diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:45-74. doi: 10.1002/dmrr.2699. No abstract available. PMID 26386266
- [Background] Breivik H, Borchgrevink PC, Allen SM, Rosseland LA, Romundstad L, Hals EK, Kvarstein G, Stubhaug A. Assessment of pain. Br J Anaesth. 2008 Jul;101(1):17-24. doi: 10.1093/bja/aen103. Epub 2008 May 16. PMID 18487245
- [Background] Meloni M, Giurato L, Izzo V, Stefanini M, Pampana E, Gandini R, Uccioli L. Long term outcomes of diabetic haemodialysis patients with critical limb ischemia and foot ulcer. Diabetes Res Clin Pract. 2016 Jun;116:117-22. doi: 10.1016/j.diabres.2016.04.030. Epub 2016 Apr 26. PMID 27321326
- [Background] Dubsky M, Jirkovska A, Bem R, Fejfarova V, Pagacova L, Nemcova A, Sixta B, Chlupac J, Peregrin JH, Sykova E, Jude EB. Comparison of the effect of stem cell therapy and percutaneous transluminal angioplasty on diabetic foot disease in patients with critical limb ischemia. Cytotherapy. 2014 Dec;16(12):1733-8. doi: 10.1016/j.jcyt.2014.08.010. Epub 2014 Oct 7. PMID 25304666
- [Background] Mustapha JA, Katzen BT, Neville RF, Lookstein RA, Zeller T, Miller LE, Jaff MR. Disease Burden and Clinical Outcomes Following Initial Diagnosis of Critical Limb Ischemia in the Medicare Population. JACC Cardiovasc Interv. 2018 May 28;11(10):1011-1012. doi: 10.1016/j.jcin.2017.12.012. No abstract available. PMID 29798766
- [Background] Klaphake S, de Leur K, Mulder PG, Ho GH, de Groot HG, Veen EJ, Verhagen HJ, van der Laan L. Mortality after major amputation in elderly patients with critical limb ischemia. Clin Interv Aging. 2017 Nov 22;12:1985-1992. doi: 10.2147/CIA.S137570. eCollection 2017. PMID 29200838
- [Background] Martini R, Andreozzi GM, Deri A, Cordova R, Zulian P, Scarpazza O, Nalin F. Amputation rate and mortality in elderly patients with critical limb ischemia not suitable for revascularization. Aging Clin Exp Res. 2012 Jun;24(3 Suppl):24-7. PMID 23160502
- [Background] Pannell M, Labuz D, Celik MO, Keye J, Batra A, Siegmund B, Machelska H. Adoptive transfer of M2 macrophages reduces neuropathic pain via opioid peptides. J Neuroinflammation. 2016 Oct 7;13(1):262. doi: 10.1186/s12974-016-0735-z. PMID 27717401
- [Background] Hasegawa T, Kosaki A, Shimizu K, Matsubara H, Mori Y, Masaki H, Toyoda N, Inoue-Shibata M, Nishikawa M, Iwasaka T. Amelioration of diabetic peripheral neuropathy by implantation of hematopoietic mononuclear cells in streptozotocin-induced diabetic rats. Exp Neurol. 2006 Jun;199(2):274-80. doi: 10.1016/j.expneurol.2005.11.001. Epub 2005 Dec 6. PMID 16337192
- [Background] Molavi B, Zafarghandi MR, Aminizadeh E, Hosseini SE, Mirzayi H, Arab L, Baharvand H, Aghdami N. Safety and Efficacy of Repeated Bone Marrow Mononuclear Cell Therapy in Patients with Critical Limb Ischemia in a Pilot Randomized Controlled Trial. Arch Iran Med. 2016 Jun;19(6):388-96. PMID 27293053
- [Background] Kang WC, Oh PC, Lee K, Ahn T, Byun K. Increasing injection frequency enhances the survival of injected bone marrow derived mesenchymal stem cells in a critical limb ischemia animal model. Korean J Physiol Pharmacol. 2016 Nov;20(6):657-667. doi: 10.4196/kjpp.2016.20.6.657. Epub 2016 Oct 28. PMID 27847443
- [Background] Fadini GP, Albiero M, Bonora BM, Avogaro A. Angiogenic Abnormalities in Diabetes Mellitus: Mechanistic and Clinical Aspects. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5431-5444. doi: 10.1210/jc.2019-00980. PMID 31211371
- [Background] Cianfarani F, Toietta G, Di Rocco G, Cesareo E, Zambruno G, Odorisio T. Diabetes impairs adipose tissue-derived stem cell function and efficiency in promoting wound healing. Wound Repair Regen. 2013 Jul-Aug;21(4):545-53. doi: 10.1111/wrr.12051. Epub 2013 Apr 29. PMID 23627689
- [Background] Rennert RC, Sorkin M, Januszyk M, Duscher D, Kosaraju R, Chung MT, Lennon J, Radiya-Dixit A, Raghvendra S, Maan ZN, Hu MS, Rajadas J, Rodrigues M, Gurtner GC. Diabetes impairs the angiogenic potential of adipose-derived stem cells by selectively depleting cellular subpopulations. Stem Cell Res Ther. 2014 Jun 18;5(3):79. doi: 10.1186/scrt468. PMID 24943716
- [Background] Navarro A, Marin S, Riol N, Carbonell-Uberos F, Minana MD. Human adipose tissue-resident monocytes exhibit an endothelial-like phenotype and display angiogenic properties. Stem Cell Res Ther. 2014 Apr 14;5(2):50. doi: 10.1186/scrt438. PMID 24731246
- [Background] Kornicka K, Houston J, Marycz K. Dysfunction of Mesenchymal Stem Cells Isolated from Metabolic Syndrome and Type 2 Diabetic Patients as Result of Oxidative Stress and Autophagy may Limit Their Potential Therapeutic Use. Stem Cell Rev Rep. 2018 Jun;14(3):337-345. doi: 10.1007/s12015-018-9809-x. PMID 29611042
- [Background] Inoue O, Usui S, Takashima SI, Nomura A, Yamaguchi K, Takeda Y, Goten C, Hamaoka T, Ootsuji H, Murai H, Kaneko S, Takamura M. Diabetes impairs the angiogenic capacity of human adipose-derived stem cells by reducing the CD271+ subpopulation in adipose tissue. Biochem Biophys Res Commun. 2019 Sep 17;517(2):369-375. doi: 10.1016/j.bbrc.2019.07.081. Epub 2019 Jul 27. PMID 31362891
- [Background] Wang SK, Green LA, Motaganahalli RL, Wilson MG, Fajardo A, Murphy MP. Rationale and design of the MarrowStim PAD Kit for the Treatment of Critical Limb Ischemia in Subjects with Severe Peripheral Arterial Disease (MOBILE) trial investigating autologous bone marrow cell therapy for critical limb ischemia. J Vasc Surg. 2017 Jun;65(6):1850-1857.e2. doi: 10.1016/j.jvs.2017.01.054. Epub 2017 Apr 5. PMID 28390770
- [Background] Hao C, Shintani S, Shimizu Y, Kondo K, Ishii M, Wu H, Murohara T. Therapeutic angiogenesis by autologous adipose-derived regenerative cells: comparison with bone marrow mononuclear cells. Am J Physiol Heart Circ Physiol. 2014 Sep 15;307(6):H869-79. doi: 10.1152/ajpheart.00310.2014. Epub 2014 Jul 25. PMID 25063790
- [Background] Kondo K, Shintani S, Shibata R, Murakami H, Murakami R, Imaizumi M, Kitagawa Y, Murohara T. Implantation of adipose-derived regenerative cells enhances ischemia-induced angiogenesis. Arterioscler Thromb Vasc Biol. 2009 Jan;29(1):61-6. doi: 10.1161/ATVBAHA.108.166496. Epub 2008 Oct 30. PMID 18974384
- [Background] Bora P, Majumdar AS. Adipose tissue-derived stromal vascular fraction in regenerative medicine: a brief review on biology and translation. Stem Cell Res Ther. 2017 Jun 15;8(1):145. doi: 10.1186/s13287-017-0598-y. PMID 28619097
- [Background] Zollino I, Campioni D, Sibilla MG, Tessari M, Malagoni AM, Zamboni P. A phase II randomized clinical trial for the treatment of recalcitrant chronic leg ulcers using centrifuged adipose tissue containing progenitor cells. Cytotherapy. 2019 Feb;21(2):200-211. doi: 10.1016/j.jcyt.2018.10.012. Epub 2018 Dec 22. PMID 30583949
- [Background] Huang P, Li S, Han M, Xiao Z, Yang R, Han ZC. Autologous transplantation of granulocyte colony-stimulating factor-mobilized peripheral blood mononuclear cells improves critical limb ischemia in diabetes. Diabetes Care. 2005 Sep;28(9):2155-60. doi: 10.2337/diacare.28.9.2155. PMID 16123483
- [Background] Fadini GP, Albiero M, Vigili de Kreutzenberg S, Boscaro E, Cappellari R, Marescotti M, Poncina N, Agostini C, Avogaro A. Diabetes impairs stem cell and proangiogenic cell mobilization in humans. Diabetes Care. 2013 Apr;36(4):943-9. doi: 10.2337/dc12-1084. Epub 2012 Oct 30. PMID 23111057
- [Background] Dong Z, Pan T, Fang Y, Wei Z, Gu S, Fang G, Liu Y, Luo Y, Liu H, Zhang T, Hu M, Guo D, Xu X, Chen B, Jiang J, Yang J, Shi Z, Zhu T, Shi Y, Liu P, Fu W. Purified CD34+ cells versus peripheral blood mononuclear cells in the treatment of angiitis-induced no-option critical limb ischaemia: 12-Month results of a prospective randomised single-blinded non-inferiority trial. EBioMedicine. 2018 Sep;35:46-57. doi: 10.1016/j.ebiom.2018.08.038. Epub 2018 Aug 29. PMID 30172703
- [Result] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Result] Reinecke H, Unrath M, Freisinger E, Bunzemeier H, Meyborg M, Luders F, Gebauer K, Roeder N, Berger K, Malyar NM. Peripheral arterial disease and critical limb ischaemia: still poor outcomes and lack of guideline adherence. Eur Heart J. 2015 Apr 14;36(15):932-8. doi: 10.1093/eurheartj/ehv006. Epub 2015 Feb 2. PMID 25650396
- [Result] Vas PRJ, Edmonds M, Kavarthapu V, Rashid H, Ahluwalia R, Pankhurst C, Papanas N. The Diabetic Foot Attack: "'Tis Too Late to Retreat!". Int J Low Extrem Wounds. 2018 Mar;17(1):7-13. doi: 10.1177/1534734618755582. Epub 2018 Feb 12. PMID 29430981